CLINICAL TRIAL: NCT00173875
Title: A Phase II Study to Evaluate the Efficacy and Safety of Iressa as a First-Line Treatment in Chemonaive Patients With Inoperable Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Iressa as a First-Line Treatment in Chemonaive Patients With Inoperable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 940107
Record Dates: First submitted 2005-09-08; First posted 2005-09-15 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2005-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Iressa
  Interventions: Drug: Iressa

INTERVENTIONS:
Drug: Iressa

SUMMARY:
The purpose of this study is to assess the overall response rate to Iressa as a first-line treatment in chemonaive patients with inoperable Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
The epidermal growth factor receptor (EGFR) is a promising target for anticancer therapy because it is expressed or highly expressed in a variety of tumors, including NSCLC.Furthermore, high levels of EGFR expression have been associated with a poor prognosis in lung cancer patients in several studies. EGFR-targeted cancer therapies are currently being developed; strategies include inhibition of the intracellular tyrosine kinase domain of the receptor by small molecules such as gefitinib (Iressa [ZD1839]; AstraZeneca, Wilmington, DE). Iressa is an orally active, selective EGFR tyrosine kinase inhibitor that blocks signal transduction pathways implicated in the proliferation and survival of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV NSCLC
* No immediate need for palliative radiotherapy and No prior chemotherapy
* age > 20 Y/O
* ECOG PS: 0 - 2
* ANC >2000
* PLT >100k
* Hb > 10
* total bilirubin < 2.0 mg/dL
* serum creatinine < 2 mg/dl
* SGPT and SGOT < 2.5 ×ULN, alkaline phosphatase < 5 ×ULN
* life expectancy >6mos.

Exclusion Criteria:

* If the patients have brain metastases or receive radiotherapy, the disease must be stable for more than 6 weeks after the last dose of radiotherapy
* 2nd malignancies
* Unable to swallow tablets
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measurements
* Pregnant or lactating patients
* Participation in other clinical trials within 30 days of study entry
* Major systemic disease which in the investigator's opinion might confound the clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the overall response rate to Iressa as a first-line treatment in chemonaive patients with inoperable Non-Small Cell Lung Cancer | 2005~2007

SECONDARY OUTCOMES:
To evaluate 1) Individual response rate 2) Time to progression 3) Overall survival (OS) at year1 4) Progression free survival (PFS) at year1 5) Toxicity | 2005~2007

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hsin Yang, M.D.,Ph.D., Principal Investigator — Department of Oncology , National Taiwan University Hospital; Ann-Lii Cheng, M.D.,Ph.D., Study Chair — Department of Oncology , National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan